CLINICAL TRIAL: NCT02636361
Title: Pharmacokinetics, Glucodynamics, Safety, and Tolerability of Multiple LY900014 Formulations
Brief Title: A Study of Various Formulations of LY900014 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 16176; I8B-FW-ITRJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-12-17; First posted 2015-12-21 (Estimated); Results first posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2016-02

CONDITIONS: Healthy
MeSH Terms: interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- LY900014 Test B (Experimental): Test formulation B: Single dose of LY900014 formulation administered subcutaneously (SC) in one of five periods
  Interventions: Drug: LY900014
- LY900014 Test A (Experimental): Test formulation B: Single dose of LY900014 formulation administered SC in one of five periods
  Interventions: Drug: LY900014
- LY900014 Test C (Experimental): Test formulation C: Single dose of LY900014 formulation administered SC in one of five periods
  Interventions: Drug: LY900014
- LY900014 Test D (Experimental): Formulation D: Single dose of LY900014 formulation administered SC in one of five periods
  Interventions: Drug: LY900014
- Insulin Lispro (Active Comparator): Reference formulation: Single dose of lispro administered SC in one of five periods
  Interventions: Drug: Insulin lispro (Humalog)

INTERVENTIONS:
Drug: LY900014 — Administered subcutaneously (SC)
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014 Test A; LY900014 Test B; LY900014 Test C; LY900014 Test D
Drug: Insulin lispro (Humalog) — Administered SC
  Other Names: Humalog; LY275585
  Arms: Insulin Lispro

SUMMARY:
This study will evaluate how quickly the body absorbs, breaks down, and gets rid of the different formulations of LY900014. This study will determine how the different formulations, when injected under the skin, will affect the blood sugar levels in the body, and how safe it is.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy male or a female (not pregnant and agreeable to take birth control measures until one month after study completion)
* Must have a body mass index (BMI) of 18.0 to 30 kilogram per square meter (kg/m²) (inclusive) at the time of study screening
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), blood and urine laboratory test results that are acceptable for the study
* Are non-smokers or have not smoked for at least 2 months prior to entering the study, and agree not to smoke (cigars, cigarettes, or pipes) or use smokeless tobacco for the duration of the study
* Have veins suitable for easy blood collection and glucose solution infusion

Exclusion Criteria:

* Have known allergies to insulin lispro or compounds related to these drugs, or any components of the study drug
* Show signs of having an infection or infectious disease at the time of study entry

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1 BDCAR: B = LY900014 Test B, D, LY900014 Test D, C = LY900014 Test C, A = LY900014 Test A, R = Reference, insulin lispro (Humalog)
- Sequence 2 ADCRB: A = LY900014 Test A, D=LY900014 Test D, C = LY900014 Test C, R = Reference, insulin lispro (Humalog), B = LY900014 Test B
- Sequence 3 ADRCB: A = LY900014 Test A, D=LY900014 Test D,R = Reference, insulin lispro (Humalog), C = LY900014 Test C, B = LY900014 Test B
- Sequence 4 BRDAC: B = LY900014 Test B,R = Reference, insulin lispro (Humalog),D=LY900014 Test D, A = LY900014 Test A,C = LY900014 Test C
- Sequence 5 RADCB: R = Reference, insulin lispro (Humalog)A = LY900014 Test A, D=LY900014 Test D, C = LY900014 Test C, B = LY900014 Test B
Period: Period 1
Arm/Group | Sequence 1 BDCAR | Sequence 2 ADCRB | Sequence 3 ADRCB | Sequence 4 BRDAC | Sequence 5 RADCB
Started | 5 | 6 | 5 | 5 | 5
Received at Least One Dose of Study Drug | 5 | 5 | 5 | 5 | 4
Completed | 5 | 5 | 5 | 5 | 4
Not Completed | 0 | 1 | 0 | 0 | 1
Period: Period 2
Arm/Group | Sequence 1 BDCAR | Sequence 2 ADCRB | Sequence 3 ADRCB | Sequence 4 BRDAC | Sequence 5 RADCB
Started | 5 | 5 | 5 | 5 | 4
Completed | 5 | 5 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 BDCAR | Sequence 2 ADCRB | Sequence 3 ADRCB | Sequence 4 BRDAC | Sequence 5 RADCB
Started | 5 | 5 | 5 | 5 | 4
Completed | 5 | 5 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1 BDCAR | Sequence 2 ADCRB | Sequence 3 ADRCB | Sequence 4 BRDAC | Sequence 5 RADCB
Started | 5 | 5 | 5 | 5 | 4
Completed | 5 | 5 | 5 | 4 | 4
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Period: Period 5
Arm/Group | Sequence 1 BDCAR | Sequence 2 ADCRB | Sequence 3 ADRCB | Sequence 4 BRDAC | Sequence 5 RADCB
Started | 5 | 5 | 5 | 4 | 4
Completed | 5 | 5 | 5 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Overall Study: All participants who received at least 1 dose of study drug.
Arm/Group | Overall Study
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 24
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 24

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under The Concentration Curve (AUC 0-30mins) of Insulin Lispro
Time Frame: Predose,5,10,15,20,25,30,35,40,45,50,55,60,70,90,120,150,180,240,300, 360 and 420 minutes postdose
Population: Participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomol per hours per liter (pmol*h/L)
Groups:
- LY900014 Test A: LY900014 Test Formulation A. Single dose of LY900014 administered subcutaneously (SC) in one of five periods.
- LY900014 Test B: LY900014 Test Formulation B. Single dose of LY900014 administered subcutaneously (SC) in one of five periods.
- LY900014 Test C: LY900014 Test Formulation C. Single dose of LY900014 administered subcutaneously (SC) in one of five periods.
- LY900014 Test D: LY900014 Test Formulation D. Single dose of LY900014 administered subcutaneously (SC) in one of five periods.
- Reference (Insulin Lispro, Humalog): A single dose of Reference (insulin lispro, Humalog) administered SC in one of five periods
Arm/Group | LY900014 Test A | LY900014 Test B | LY900014 Test C | LY900014 Test D | Reference (Insulin Lispro, Humalog)
Number analyzed (Participants) | 24 | 24 | 23 | 24 | 24
picomol per hours per liter (pmol*h/L) | 245 (65) | 295 (54) | 251 (45) | 253 (56) | 120 (101)

2. Secondary Outcome: Total Amount of Glucose Infused (Gtot) Over the Duration of Clamp
Time Frame: Predose, every 2.5 minutes for 30 minutes, then every 5 min until 120 minutes, then every 10 minutes until 300 minutes, then every 20 minutes until 480 minutes.
Population: All participants who received at least 1 dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams (mg)
Groups:
- LY900014 Test A: LY900014 Test Formulation A: Single dose of LY900014 formulation administered subcutaneously (SC) in one of five periods.
- LY900014 Test D: LY900014 Test Formulation B. Single dose of LY900014 administered subcutaneously (SC) in one of five periods.
Arm/Group | LY900014 Test A | LY900014 Test B | LY900014 Test C | LY900014 Test D | Reference (Insulin Lispro, Humalog)
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
milligrams (mg) | 84300 (35) | 91100 (35) | 91300 (27) | 88700 (34) | 85400 (32)

ADVERSE EVENTS:
Groups:
- Reference (Insulin Lispro, Humalog): Reference formulation: Single dose of lispro administered SC in one of five periods
- LY900014 Test A: Test formulation A: Single dose of LY900014 formulation administered subcutaneously (SC) in one of five periods
- LY900014 Test C: Test formulation C: Single dose of LY900014 formulation administered subcutaneously (SC) in one of five periods
- LY900014 Test D: Test formulation D: Single dose of LY900014 formulation administered subcutaneously (SC) in one of five periods
Arm/Group | Reference (Insulin Lispro, Humalog) | LY900014 Test A | LY900014 Test B | LY900014 Test C | LY900014 Test D
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 1/24 | 0/24 | 2/24 | 1/23 | 3/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reference (Insulin Lispro, Humalog) (N=24) | LY900014 Test A (N=24) | LY900014 Test B (N=24) | LY900014 Test C (N=23) | LY900014 Test D (N=24)
Catheter site related reaction (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days